CLINICAL TRIAL: NCT04306510
Title: A Phase 4 Safety Study Assessing the Adverse Events Occurring Within One Day of TEGSEDI Administration in Patients With Polyneuropathy of Hereditary Transthyretin-mediated Amyloidosis (hATTR-PN)
Brief Title: A Study to Characterize Adverse Events Occurring Within One Day of TEGSEDI Administration to Adult Participants With hATTR-PN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawal of TEGSEDI from sale was not related to any safety issues.
Sponsor: Akcea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TEG4004
Record Dates: First submitted 2020-02-07; First posted 2020-03-13 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Hereditary Transthyretin Amyloidosis With Polyneuropthy
Keywords: Hereditary Transthyretin Amyloidosis; hATTR-PN; hATTR; Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis | interventions — Inotersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TEGSEDI (Experimental): Participants received TEGSEDI 284 milligrams (mg), subcutaneously (SC) once weekly, as prescribed by their physician per the product label.
  Interventions: Drug: TEGSEDI

INTERVENTIONS:
Drug: TEGSEDI — SC injection.
  Other Names: Inotersen

SUMMARY:
The objective of the study was to characterize adverse events (AEs) occurring within one day of TEGSEDI administration to adult participants with hATTR-PN overall and in individual participants with respect to time course of AE onset, vital sign changes, preventive measures, treatment required, risk factors, and subsequent adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Satisfy one of the following:

   1. United States (US) Participants: Adult participants (≥ 18 years old) diagnosed with hATTR-PN and prescribed TEGSEDI according to the United States Prescribing Information (USPI).
   2. Canadian participants: Adult participants (≥ 18 years old) diagnosed with stage 1 or stage 2 hATTR-PN and prescribed TEGSEDI according to the Canadian Product Monograph (CPM).
2. Must have given written informed consent for participation in this study.
3. Must provide access to their previous medical records.
4. Are about to initiate or have recently initiated treatment with TEGSEDI and have not received more than 9 doses in total.
5. Be willing to complete required testing and report any AEs and/or changes in medications.
6. Satisfy one of the following:

   1. Females: Non-pregnant and non-lactating; abstinent, or if engaged in sexual relations of childbearing potential, participant is using an acceptable contraceptive method from time of signing the informed consent form (ICF) until 13 weeks after the last dose of TEGSEDI administration
   2. Males: Abstinent or if engaged in sexual relations with a female of childbearing potential, participant is utilizing an acceptable contraceptive method from the time of signing the ICF until 13 weeks after the last dose of TEGSEDI administration

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Study Center, Rosedale, New York, United States
- Study Center, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 2 clinical sites in the United States of America (USA) and Canada from 21 January 2021 to 20 March 2024.
Pre-assignment Details: A total of 8 participants with polyneuropathy of hereditary transthyretin-mediated amyloidosis (hATTR-PN) were screened for the study, of which 7 participants were treated with TEGSEDI. The 8th participant was enrolled after the sponsor had notified the sites about the study close-out activities, therefore only 7 participants were included in the study.
Period: Overall Study
Arm/Group | TEGSEDI
Started | 8
Completed | 6
Not Completed | 2
Not completed — Voluntarily withdrawal | 1
Not completed — Enrolled but Not Treated | 1

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least 1 dose of TEGSEDI while enrolled in this study protocol.
Groups:
- TEGSEDI: Participants with hATTR-PN received TEGSEDI 284 mg, SC once weekly, as prescribed by their physician per the product label.
Arm/Group | TEGSEDI
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 4
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incident, Onset and Duration of Treatment Emergent Adverse Events (TEAEs) Occurring Within 24 Hours of Each TEGSEDI Administration
Description: An adverse event (AE) is defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of medicinal product, whether or not the AE is considered related to the medicinal product. TEAEs are defined as AEs with an onset date/time on or after the date/time of the first on study administration of TEGSEDI.
Time Frame: Up to 2 years (24 hours post each TEGSEDI injection)
Population: The evaluable set included participants in the safety set having at least 1 post-dose assessment.
Measure: Count of Participants; unit: Participants
Groups:
- TEGSEDI: Participants received TEGSEDI 284 mg, SC once weekly, as prescribed by their physician per the product label.
Arm/Group | TEGSEDI
Number analyzed (Participants) | 7
Participants | 3

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs including body temperature, heart rate, respiratory rate, and systolic/diastolic blood pressure (BP).
Time Frame: Up to 2 years (24 hours post each TEGSEDI injection)
Population: The evaluable set included participants in the safety set having at least 1 post-dose assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | TEGSEDI
Number analyzed (Participants) | 7
Participants | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Cytokine Levels and Inflammatory Markers
Description: Cytokines and inflammatory markers including the following parameters: Immunoglobulin (Ig)E, IgG, IgM, C-reactive protein, erythrocyte sedimentation rate, interferon-alpha, interferon beta, chemokines (macrophage inflammatory protein-1a and membrane cofactor protein-1, granulocyte-macrophage colony-stimulating factor, Interleukin (IL)-1alpha (α), IL-1 beta (β), IL-6, IL-8, IL-12, and tumor necrosis factor-α.
Time Frame: Up to 2 years (24 hours post each TEGSEDI injection)
Population: The evaluable set included participants in the safety set having at least 1 post-dose assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | TEGSEDI
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years (24 hours post each TEGSEDI injection)
Description: The evaluable set included participants in the safety set having at least 1 post-dose assessment.
Arm/Group | TEGSEDI
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEGSEDI (N=7)
Chills (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site discomfort (General disorders) | 1
Injection site pain (General disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This study was subject to limitations due to the rarity of hATTR-PN, which limits the enrollment of potentially eligible patients. Additionally, the availability of concurrent clinical trials and newer therapies targeting the same patient population further complicated efforts to achieve the planned enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT04306510/Prot_SAP_000.pdf